CLINICAL TRIAL: NCT00393744
Title: A Phase III, Open, Randomised, Multicentre Study Comparing the Efficacy and Safety of Pristinamycin, at Dosages of 50 mg/kg/d in 2 Doses for Children, and 1g Twice Daily in Adults for 4 Days Versus Amoxicillin at a Dosage of 50 mg/kg/d in 2 Doses in Children and 1 g Twice Daily in Adults for 6 Days, Consumed Orally, in the Treatment of Tonsillitis Induced by Group-A Beta-Haemolytic Streptococcus in Patients Aged Between 6 and 25 Years.
Brief Title: Efficacy Study of Pristinamycin Versus Amoxicillin to Treat Tonsillitis Induced by Streptococcus in Children
Acronym: PRI-angine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIST_L_01683; EudraCT #: 2006-002127-16
Record Dates: First submitted 2006-10-27; First posted 2006-10-30 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-03

CONDITIONS: Tonsillitis
MeSH Terms: conditions — Tonsillitis | interventions — Pristinamycin; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: pristinamycin
- 2 (Active Comparator)
  Interventions: Drug: amoxicillin

INTERVENTIONS:
Drug: pristinamycin — 50 mg/kg/d in 2 doses for children, and 1g twice daily in adults for 4 days
  Arms: 1
Drug: amoxicillin — 50 mg/kg/d in 2 doses in children and 1 g twice daily in adults for 6 days
  Arms: 2

SUMMARY:
The primary objective of this study is to demonstrate the non-inferiority, at the assessment visit (V3 (D10/D14)), in terms of bacteriological efficacy of pristinamycin (PRI) administered for 4 days versus amoxicillin (AMX) administered for 6 days in the treatment of tonsillitis caused by GAS, in subjects aged between 6 and 25 in the per protocol (PP) group.

ELIGIBILITY:
Inclusion Criteria:

* subjects of both sexes
* aged between 6 and 25 years,
* weight : ≥ 20kg
* with suspected GAS-induced tonsillitis (erythema and/or exudate of the pharynx and/or tonsils with oropharyngeal pain and/or odynophagia, fever ³ 38°C, appreciable satellite adenopathy)
* confirmation by positive RDT
* provision of throat swabs for culture
* ability to swallow tablets

Exclusion Criteria:

* Related to the study disease:

  * suspected viral infection (concomitant dysphonia, cough, conjunctivitis, rhinitis)
  * adenophlegmon, peritonsillar abscesses.
* Related to the study treatment:

  * known or suspected allergy to beta-lactamines (penicillin, cephalosporin)
  * suspected infectious mononucleosis (increased risk of skin disorders)
  * phenylketonuria (due to the presence of aspartame)
  * congenital galactosaemia, glucose/galactose malabsorption syndrome, lactase deficiency (due to the presence of lactose, in powder or suspension form)
  * allergy to pristinamycin and/or virginiamycin
  * history of pustular rash with pristinamycin
  * hypersensitivity or gluten intolerant (due to the presence of wheat starch)
  * ongoing treatment with cyclosporine, methotrexate, colchicine, allopurinol, tacrolimus or oral anticoagulants.
* Related to previous treatment:

  * subjects receiving antibiotic therapy in the month prior to inclusion, except for azithromycin, for which the exclusion period is 3 months.
  * subjects on short-term corticosteroids. Subjects on long-term corticosteroids initiated before the start of the study and taken at a controlled dosage may be included.
* Related to subjects:

  * breast-feeding women
  * women either pregnant or attempting to conceive
  * subjects likely, during the course of the study to receive treatments prohibited by the protocol
  * treatment with other investigational drugs in the 4 weeks prior to inclusion in the study
  * immunodepression, clinically significant endocrine disease, cardiovascular disease, neurological disease, or any other marked diseases resulting in complications in performance of the study or interpretation of the study data
  * known hepatic impairment
  * known renal impairment (creatinine clearance < 30 ml/minute)
  * cancer, blood dyscrasias
  * previous history of drug or alcohol abuse.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 395 (Actual)
Dates: Start 2006-10; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
bacterial eradication | at V3

SECONDARY OUTCOMES:
adverse events | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Marie SEBILLE, Dr, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France